CLINICAL TRIAL: NCT03827850
Title: A Phase II Trial to Evaluate Efficacy and Safety of Erdafitinib in Patients With Advanced Non Small Cell Lung Carcinoma (NSCLC) Harboring Fibroblast Growth Factor Receptor (FGFR) Genetic Alterations After Relapse of Standard Therapy.
Brief Title: FGFR Inhibitor in FGFR Dysregulated Cancer
Acronym: FIND
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study-related difficulties faced with patient enrolment, no safety-related reasons
Sponsor: Lung Cancer Group Cologne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-3254; 2018-000399-13 (EudraCT Number)
Record Dates: First submitted 2019-01-22; First posted 2019-02-04 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Lung Cancer; NSCLC; Pulmonary Neoplasm; Squamous Cell Lung Cancer; NSCLC Stage IV
Keywords: sqNSCLC; FGFR Mutations
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — erdafitinib

STUDY DESIGN:
Intervention Model Description: Patients with NSCLC and FGFR alteration with high evidence on oncogenic transformation according to FIND molecular board will be included to cohort 1 (FGFR translocated NSCLC patients) and cohort 2 (FGFR mutated NSCLC patients). Patients with NSCLC and FGFR alterations without enough evidence (intermediate / low evidence according to FIND molecular tumor board) for recruitment into cohorts 1 or 2, will be treated in cohort 3. Overall response rate under Erdafitinib treatment will be the primary endpoint.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 FGFR trans (Active Comparator): Cohort 1: Activating (high confidence) FGFR translocations (max. 15 patients) under daily Erdaifitinib treatment
  Interventions: Drug: ERDAFITINIB
- Cohort 2 FGFR mut (Active Comparator): Cohort 2: Activating (high confidence) hotspot FGFR mutations (max. 15 patients) under daily Erdafitinib treatment
  Interventions: Drug: ERDAFITINIB
- Cohort 3 FGFR other (Active Comparator): Cohort 3: Activating (low confidence) FGFR alteration (max. 20 patients)
  Interventions: Drug: ERDAFITINIB

INTERVENTIONS:
Drug: ERDAFITINIB — Daily in a range from 3 mg to 9 mg
  Other Names: JNJ -42756493; WHO NUMBER 10147

SUMMARY:
In the FIND trial, Non Small Cell Lung Carcinoma (NSCLC) patients with Fibroblast Growth Factor Receptor (FGFR) genetic alteration will be treated with the selective FGFR1-4 inhibitor erdafitinib. Archival samples, fresh frozen tumor samples and blood for circulating tumor DNA (ctDNA) will be collected before treatment. Patients will be treated until disease progression or unacceptable toxicity. In case of progression, fresh frozen tumor biopsies and ctDNA analyses will be performed to assess resistance mechanisms. The primary objective of the trial is to analyze the efficacy of erdafitinib in NSCLC patients with FGFR genetic alterations. NSCLC patient number will be based on a statistical hypothesis aiming at increasing the response rate comparing to chemotherapy/immunotherapy after standard treatment.

DETAILED DESCRIPTION:
Downstream signaling of fibroblast growth factor receptors 1-4 (FGFR 1-4) regulates cell proliferation, migration, differentiation and survival in healthy cells. Genetic alterations (amplifications, point-mutations and translocations) in FGFR1-4 genes cause altered signaling and oncogenic transformation. FGFR-alterations with sensitivity to kinase inhibition have been identified in a variety of tumors such as breast-, bladder- and endometrial-cancer, squamous cell lung and head and neck cancer, cholangiocarcinoma and glioblastoma.

First-in-man/phase-I clinical trials with erdafitinib and BGJ398 - both selective FGFR inhibitors - enrolled patients with any genetic alterations in FGFR. The trials showed clinical responses with differences according to the type of FGFR alterations and histological subtypes. In the BGJ398 trial, the partial response rate was 11% (4/36) in patients with FGFR1 amplified squamous NSCLC (sqNSCLC) and 38% (3/8) in patients with FGFR3-mutant bladder cancer. No PR was observed in patients with FGFR1/2 amplified (n=25) and FGFR3 mutant (n=1) breast cancer. All patients with FGFR2-translocated (n=2) and FGFR2-mutated cholangiocarcinoma (n=1) showed reduced tumor burden of 20% and 10%, respectively. In the erdafitinib trial, 5 partial responses were seen in FGFR translocated tumors: 3/8 (37.5%) patients with urothelial carcinoma, 1/3 (33%) patients with glioblastoma and 1 patient with endometrial cancer reached PR. Summing up the results of the phase-I trials, the inhibition of FGFR downstream pathways in FGFR translocated and mutated solid tumors exerted clinical activity. Thus, focusing treatment with FGFR inhibitors on FGFR mutated and translocated solid tumors may increase response rates, progression free and overall survival in these tumors with otherwise adverse prognosis.

In NSCLC patients without druggable alterations in genes as EGFR, ALK or ROS1 and without high PD-L1 (Programmed cell death 1 ligand 1) expression, prognosis remains adverse with a median survival time of about 18 months. Particularly in sqNSCLC, only few driver mutations have been identified yet. Of these, solely mutations of the KRAS gene (although observed at low frequency in sqNSCLC) were explored in large clinical studies targeting KRAS downstream signaling with no survival benefit comparing to chemotherapy. Immunotherapy with PD-1 antibodies such as nivolumab and pembrolizumab showed benefit in patients with high PD-L1 expression mainly.

The frequency of somatic FGFR1-3 mutations in lung cancer is about 4% (Helsten et al., 2016). Translocations occur with a similar frequency of about 4% in lung cancer. Multiple of these FGFR alterations are shown to have oncogenic potential as demonstrated in multiple in vitro, in vivo and first-in-man studies.

Preclinical models in NSCLC cell lines and xenografts showed oncogenic activity of FGFR2/3 mutations with consecutive sensitivity to FGFR inhibitors. Similarly, FGFR3-TACC translocation exerted kinase activation in sqNSCLC cell lines and other tumor types. Furthermore, patient derived FGFR3-fusion lung xenograft model showed responses to FGFR targeted treatment.

In summary, on the basis of genetically and phenotypically validated cell-line panels, in vivo and particularly on the basis of clinical data, there is strong evidence for a clinical benefit from FGFR inhibition for patients with FGFR altered NSCLC.

The primary objective of the trial is to analyze the efficacy of erdafitinib in NSCLC patients with FGFR genetic alterations. NSCLC patient number will be based on a statistical hypothesis aiming at increasing the response rate comparing to chemotherapy/immunotherapy after standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Stage IIIB/IV NSCLC patients with activating FGFR alteration after the failure on any prior line of standard treatment, or in the opinion of the investigator no effective standard therapy exists, is appropriate, tolerated or is considered equivalent to study treatment
* Activating FGFR alteration as approved by FIND Molecular Board
* Must sign an informed consent form (ICF) (or their legally acceptable representative must sign) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study.
* ECOG performance status score 0, 1, or 2.
* Clinical laboratory values and cardiovascular measurements at screening as defined in protocol
* Disease measurable per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) for cohort 1 and 2. or evaluable disease.
* A woman of childbearing potential who is sexually active must have a negative pregnancy test (human chorionic gonadotropin [hCG]) at Screening (urine or serum, minimum sensitivity 25 IU/L or equivalent units of b-HCG) within 24 hours prior to the start of erdafitinib
* Women of childbearing potential (WOCBP) and men who are sexually active with WOCBP must use appropriate method(s) of contraception with a failure rate of less than 1% per year before study entry, during the study and until 5 months after taking the last dose of study drug. And other Criteria

Exclusion Criteria:

* Pathogenic somatic alterations in the following genes: EGFR, BRAF, ALK, ROS1 and NTRK (Please note that molecular testing might be reduced in heavy smokers with NSCLC)
* Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days prior to recruitment
* Treatment with small molecules or chemotherapy within 7 days prior C1D1
* Treatment with monoclonal antibodies within 28 days prior C1D1 if related to the underlying malignancy
* Any other history of ongoing malignancy that would potentially interfere with the interpretation of erdafitinib efficacy
* Symptomatic central nervous system metastases.
* Received prior FGFR inhibitor treatment or if the patient has known allergies, hypersensitivity, or intolerance to erdafitinib or its excipients
* Any corneal or retinal abnormality likely to increase the risk of eye toxicity, i.e.:
* History of or current evidence of CeSR or retinal vascular occlusion (RVO)
* Active wet, age-related macular degeneration (AMD)
* Diabetic retinopathy with macular edema (non-proliferative)
* Uncontrolled glaucoma (per local standard of care)
* Corneal pathology such as keratitis, keratoconjunctivitis, keratopathy, corneal abrasion, inflammation or ulceration.
* Has persistent phosphate level >ULN during screening (on 2 consecutive assessments at least 1 week apart, within 14 days prior to Cycle 1 Day 1) and despite medical management
* Has a history of or current uncontrolled cardiovascular disease as defined in protocol
* Known human immunodeficiency virus (HIV) infection, testing is mandatory (a-HIV 1/2)
* Patients with acute or chronic Hepatitis B infection (tests should include assessment of HBsAg and HBc IgG antibody. If one parameter is positive, determine HBV-DNA to confirm acute infection. Patients with positive results for HBsAg and/or HBV-DNA are considered positive for acute or chronic infection.
* Patients with acute or chronic Hepatitis C infection (determine HCV-RNA. Patients with positive result for HCV-RNA are considered positive for acute or chronic infection).
* Has not recovered from reversible toxicity of prior anticancer therapy (except toxicities which are not clinically significant such as alopecia, skin discoloration, Grade 1 neuropathy, Grade 1-2 hearing loss)
* Has impaired wound healing capacity defined as skin/decubitus ulcers, chronic leg ulcers, known gastric ulcers, or unhealed incisions
* Major surgery within 2 weeks of the first dose, or will not have fully recovered from surgery, or has surgery planned during the time the patient is expected to participate in the study or within 2 weeks after the last dose of study drug administration. (patients with planned surgical procedures to be conducted under local anesthesia may participate).
* Any serious underlying medical condition, such as:

  * Evidence of serious active viral, bacterial, or uncontrolled systemic fungal infection requiring current systemic treatment
  * Psychiatric conditions (eg, alcohol or drug abuse), dementia, or altered mental status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-14 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | 3 years
  Overall response rate (ORR) per RECIST 1.1 under erdafitinib treatment in sqNSCLC with genetic alteration in FGFR

SECONDARY OUTCOMES:
number of adverse events per patient | 3 years
  assessment of adverse events according to CTC-AE
time length of progression free survival | 3 years
  assessment of progression free survival
time length of overall survival | 3 years
  assessment of overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Nogova, MD, Principal Investigator — University Clinic Cologne
Locations (11):
- Germany (11):
  - Asklepios Klinik München Gauting, Gauting, Bavaria
  - Uniklinik Frankfurt, Frankfurt am Main, Hesse
  - Städtisches Klinikum Braunschweig, Braunschweig, Lower Saxony
  - Pius Hospital Oldenburg, Oldenburg, Lower Saxony
  - Uniklinik RWTH Aachen - Klinik für Hämotologie, Onkologie, Aachen, North Rhine-Westphalia
  - University Hospital of Cologne, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Würzburg Comprehensive Cancer center, Würzburg, North Rhine-Westphalia
  - Uniklinik Carl Gustav Carus Dresden, Dresden, Saxony
  - Evangelische Lungenklink Berlin, Berlin
  - Universitätsklinik Freiburg, Freiburg im Breisgau
  - Universitätsklinik des Saarlandes Homburg, Homburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nogova L, Sequist LV, Perez Garcia JM, Andre F, Delord JP, Hidalgo M, Schellens JH, Cassier PA, Camidge DR, Schuler M, Vaishampayan U, Burris H, Tian GG, Campone M, Wainberg ZA, Lim WT, LoRusso P, Shapiro GI, Parker K, Chen X, Choudhury S, Ringeisen F, Graus-Porta D, Porter D, Isaacs R, Buettner R, Wolf J. Evaluation of BGJ398, a Fibroblast Growth Factor Receptor 1-3 Kinase Inhibitor, in Patients With Advanced Solid Tumors Harboring Genetic Alterations in Fibroblast Growth Factor Receptors: Results of a Global Phase I, Dose-Escalation and Dose-Expansion Study. J Clin Oncol. 2017 Jan 10;35(2):157-165. doi: 10.1200/JCO.2016.67.2048. Epub 2016 Nov 21. PMID 27870574
- [Background] Hierro C, Rodon J, Tabernero J. Fibroblast Growth Factor (FGF) Receptor/FGF Inhibitors: Novel Targets and Strategies for Optimization of Response of Solid Tumors. Semin Oncol. 2015 Dec;42(6):801-19. doi: 10.1053/j.seminoncol.2015.09.027. Epub 2015 Sep 24. PMID 26615127
- [Background] Schildhaus HU, Nogova L, Wolf J, Buettner R. FGFR1 amplifications in squamous cell carcinomas of the lung: diagnostic and therapeutic implications. Transl Lung Cancer Res. 2013 Apr;2(2):92-100. doi: 10.3978/j.issn.2218-6751.2013.03.03. PMID 25806220